CLINICAL TRIAL: NCT03268018
Title: ModificatiOn and Treatment of stenoseD Calcified inFrainguinal Lesions With Laser atherectomY in a Pilot Study
Acronym: MODIFY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D034698
Record Dates: First submitted 2017-07-11; First posted 2017-08-31 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-09

CONDITIONS: Peripheral Arterial Disease
Keywords: calcium; peripheral arterial disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other)
  Interventions: Device: Laser induced pressure wave calcium modification

INTERVENTIONS:
Device: Laser induced pressure wave calcium modification — A calcium atherectomy and modification solution in patients with balloon resistant calcified lesions in infrainguinal disease. The intent is to both debulk and modify the vessel to restore blood flow, improve vessel compliance and drive better outcomes
  Other Names: Laser atherectomy

SUMMARY:
The MODIFY Pilot clinical study in Europe looks to evaluate acute and procedural outcomes using a new calcium atherectomy and modification solution in patients with balloon resistant calcified lesions in infrainguinal disease. The intent is to both debulk and modify the vessel to restore blood flow, improve vessel compliance and drive better outcomes. The MODIFY Pilot study will evaluate safety and performance measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ≥ 18 years
2. Patient agrees to participate and comply with the protocol by signing an Ethics Committee approved consent form
3. Peripheral arterial disease with a documented Rutherford Class 2-5 and

   1. a resting ankle-brachial index (ABI) of <0.9 or an abnormal exercise ABI (<0.75) if resting ABI is normal. Patient with incompressible arteries (ABI >1.2) must have a toe brachial index (TBI) <0.7 in target limb;
   2. or a previous intervention to the target vessels with reoccurrence of symptoms
4. Balloon resistant calcific lesion apparent on angiogram by inability to dilate lesion to less than 50% diameter stenosis (DS)
5. Lesion to include fluoroscopic evidence of calcification: 1) on parallel sides of the vessel and 2) extending greater than 1 cm in length
6. De novo or restenotic lesion of the SFA, popliteal or infrapopliteal artery
7. Minimum reference vessel diameter (RVD) of 2.5mm
8. Minimum target lesion length of ≥ 5cm
9. At least one patent (<50% stenosed) runoff vessel to the foot

Exclusion Criteria:

1. Patient is pregnant or breast feeding (Female subjects of childbearing potential must have negative serum pregnancy test 7 days prior to treatment)
2. Life expectancy < 12 months
3. Cerebrovascular accident < 60 days prior to procedure
4. Myocardial infarction < 60 days prior to procedure
5. Known contraindication to aspirin, antiplatelet/anti-coagulant therapies required for procedure/follow up
6. Known allergy to contrast media that cannot adequately be pre-medicated prior to study procedure
7. Uncontrolled hypercoagulability or history of HIT or HITT syndrome
8. Serum creatinine ≥ 2.5 mg/dL tested within a week prior to procedure
9. Patient is simultaneously participating in another investigational drug or device study that will interfere with the 30 day Safety Endpoint
10. Patient is not eligible for bypass surgery or endovascular intervention
11. Planned major amputation
12. Planned or predicted cardiovascular surgical or interventional procedures prior to completion of the 30-day follow-up (including, but not limited to aortic, renal, cardiac, carotid, contralateral femoropopliteal, and contralateral below the knee
13. Lesion located within a stent or endograft
14. Ipsilateral and/or contralateral iliac (or common femoral) artery stenosis ≥ 50% DS that is not successfully treated prior to index procedure
15. Target lesion could not be crossed with the guidewire or support catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-03-18 (Actual)

PRIMARY OUTCOMES:
Primary performance defined as minimum lumen diameter measured pre-laser atherectomy and post-calcium modification as well as the ability to dilate a previously balloon resistant lesion after calcium modification procedure | Index procedure
  Minimum Lumen Diameter (MLD) measured pre-laser atherectomy and post-calcium modification, as measured by angiography and QVA.
  The ability to dilate a previously balloon resistant lesion after calcium modification procedure with low pressure balloon inflation.
Primary safety as defined as major adverse event (MAE) composite of all cause death, target vessel revascularization and major amputation of the target limb. | 30 days
  Safety outcome through 30-day follow-up (MAE composite):
  All cause death Target vessel revascularization (TVR) Major amputation of target limb

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - AZ Sint Blasius, Dendermonde

IPD SHARING:
Plan to Share IPD: No